CLINICAL TRIAL: NCT00000686
Title: A Phase I Safety Study of BMY-27857 (2',3'-Dideoxy-2',3'-Didehydrothymidine [d4T]) Administered Four Times Daily to AZT-Intolerant Patients With AIDS or AIDS-Related Complex
Brief Title: A Study of d4T in Patients With AIDS or AIDS-Related Complex Who Cannot Take AZT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 111; AI455-004
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 1999-05

CONDITIONS: HIV Infections
Keywords: Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Stavudine

INTERVENTIONS:
Drug: Stavudine

SUMMARY:
To determine the safety and maximum tolerated dose (MTD) of 2',3'-dideoxy-2',3'-didehydrothymidine (d4T) administered to patients with AIDS or AIDS related complex (ARC) who are intolerant of zidovudine (AZT). The study also begins an assessment of the effectiveness of d4T therapy on HIV replication, on plasma levels of p24 antigen, and clinical or immunologic parameters associated with AIDS.

Of the methods that are being evaluated to treat HIV-infected individuals, AZT has produced the best results to date. Toxic effects in approximately 50 percent of patients receiving AZT may limit its usefulness for prolonged treatment. Long-term treatment may be necessary to prevent progression of early stage HIV infection to AIDS and to prevent secondary transmission. Other drugs that may be equally or more effective than AZT and useful in the long- term treatment of HIV infection must be developed and evaluated. Test-tube and animal studies of d4T show that the drug can inhibit replication (reproduction) of HIV at concentrations similar to concentrations of AZT that have anti-HIV activity. These studies also indicate that the drug may stay in the bloodstream longer than AZT. Thus, it may be possible for the drug to be as effective as AZT when taken less frequently than AZT. It also may have a less disturbing effect on other body functions (such as thymidine metabolism).

DETAILED DESCRIPTION:
Of the methods that are being evaluated to treat HIV-infected individuals, AZT has produced the best results to date. Toxic effects in approximately 50 percent of patients receiving AZT may limit its usefulness for prolonged treatment. Long-term treatment may be necessary to prevent progression of early stage HIV infection to AIDS and to prevent secondary transmission. Other drugs that may be equally or more effective than AZT and useful in the long- term treatment of HIV infection must be developed and evaluated. Test-tube and animal studies of d4T show that the drug can inhibit replication (reproduction) of HIV at concentrations similar to concentrations of AZT that have anti-HIV activity. These studies also indicate that the drug may stay in the bloodstream longer than AZT. Thus, it may be possible for the drug to be as effective as AZT when taken less frequently than AZT. It also may have a less disturbing effect on other body functions (such as thymidine metabolism).

Five patients are enrolled at each dose level and receive d4T for 10 weeks at their initial dose level. Escalation to the next higher dose level, using a different group of five patients, occurs after three patients in the preceding group have successfully completed at least 3 weeks of oral dosing.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Diagnosis of AIDS or AIDS related complex (ARC).
* Previous intolerance to daily doses of up to 1200 mg of zidovudine (AZT) demonstrated by a decrease in hemoglobin levels of 2 - 8.5 g/dl or AZT-related depression of neutrophils of 200 - 750 cells/mm3.
* Ability to provide informed consent.

Prior Medication:

Allowed:

* Zidovudine (AZT).

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* AIDS-defining opportunistic infection on enrollment.
* Intractable diarrhea.
* History of seizures within past 2 years or currently requiring anticonvulsants for control.
* Any other clinical conditions or prior therapy which in the opinion of the investigator would make the patient unsuitable for study or unable to comply with the dosing requirements.

Concurrent Medication:

Excluded:

* Systemic maintenance or chemoprophylaxis for opportunistic infection (includes dapsone, acyclovir).
* Systemic therapy with this or any other antiretroviral drug (except zidovudine (AZT)) or investigational drug.
* Ribavirin.
* Cytotoxic anticancer therapy.
* Any agent known as a potent inducer or inhibitor of drug-metabolizing enzymes (includes rifampin and barbiturates).
* Trimethoprim / sulfamethoxazole (TMP / SMX).

Patients with the following are excluded:

* AIDS-defining opportunistic infection on enrollment.
* Intractable diarrhea.
* History of seizures within past 2 years or currently requiring anticonvulsants for control.
* Any other clinical conditions or prior therapy which in the opinion of the investigator would make the patient unsuitable for study or unable to comply with the dosing requirements.

Prior Medication:

Excluded within 2 weeks of study entry:

* Any agent known as a potent inducer or inhibitor of drug-metabolizing enzymes (includes rifampin and barbiturates).

Excluded within 1 month of study entry:

* Systemic therapy with this or any other antiretroviral drug (except zidovudine (AZT)) or investigational drug.

Excluded within 3 months of study entry:

* Ribavirin.
* Cytotoxic anticancer therapy.

Active alcohol or drug abuse sufficient in investigator's opinion to prevent adequate compliance with study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell Univ Med Ctr, New York, New York, United States

REFERENCES:
- [Background] Browne MJ, Mayer KH, Chafee SB, Dudley MN, Posner MR, Steinberg SM, Graham KK, Geletko SM, Zinner SH, Denman SL, et al. 2',3'-didehydro-3'-deoxythymidine (d4T) in patients with AIDS or AIDS-related complex: a phase I trial. J Infect Dis. 1993 Jan;167(1):21-9. doi: 10.1093/infdis/167.1.21. PMID 8093363